CLINICAL TRIAL: NCT06028568
Title: The Reliability and Validity of Perioperative Cognitive Test Network Platform for Monitoring Perioperative Neurocognitive Function Changes in Patients Undergoing Surgery
Brief Title: The Reliability and Validity of Perioperative Cognitive Test Network Platform for Monitoring Neurocognitive Changes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20232188-C-1
Record Dates: First submitted 2023-07-07; First posted 2023-09-08 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-06

CONDITIONS: Perioperative Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elderly patients undergoing surgery: Older than or equal to 65 years of age; patients who intend to undergo major abdominal surgery under general anesthesia (grade 3-4 surgery based on surgical grade)
- Elderly healthy volunteers: Age-and sex-matched community population

SUMMARY:
This study aimed to analyze the reliability and validity of the results of the new designed perioperative cognitive test network platform, and to judge the reliability and scientific nature of the perioperative cognitive test. And then to explore whether the perioperative cognitive test network platform can be used to evaluate the changes of perioperative cognitive function of patients.

DETAILED DESCRIPTION:
Two cohorts of elderly healthy volunteers and elderly patients undergoing abdominal surgery will be included in this study. The cognitive function of the patients was tested one day before and seven days after operation. Healthy volunteers had two cognitive function tests at the same interval. The normality test is used to evaluate whether the test results accord with the normal distribution. The internal consistency of the test was evaluated by calculating the Cronbach coefficient, the content validity was evaluated by experts and the content validity index was calculated, and the construct validity of the test was evaluated by exploratory factor analysis and confirmatory factor analysis. The validity of the test was evaluated by calculating the effect scale.

ELIGIBILITY:
Inclusion Criteria:

* Age over 65
* Scheduled for abdominal surgery under general anesthesia (grade 3-4 surgery based on surgical grade)
* Informed consent has been obtained
* Healthy volunteer groups are listed as age-and sex-matched community groups

Exclusion Criteria:

* Unable to follow instruction and finish the firtst procedure
* Has severe visual or auditory problems
* History of drug or alcohol abuse (drinking more than 5U daily in the past 3 months, 1U equals 10ml or 8g pure alcohol, equivalent to >50 liquor over 100ml, two two
* Are diagnosed neuropsychological disease that needs treatment
* Clear history of severe cerebrovascular diseases (including cerebral hemorrhage and cerebral infarction), Parkinson's syndrome, schizophrenia, bipolar disorder, depression, dementia, Alzheimer's disease, etc
* Severe head trauma, carbon monoxide poisoning and other loss of consciousness more than 30 minutes
* MMSE score ≤23
* Participated this study or being participating other clinical research

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study will include two groups: elderly healthy volunteers and elderly patients undergoing abdominal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Reliability | Baseline Test：1 day before operation, Second Test: Day 7 after operation
  Cronbach's alpha is used to assess the reliability and the internal consistency of this Cognitive test.
  Cronbach's alpha value >0.7 indicating the reliability of the test is acceptable.
Validity | Baseline Test：1 day before operation, Second Test: Day 7 after operation
  Content validity, Construct validity and Responsiveness analysis are used to evaluate the validity of the cognitive test.
  The item-content validity index (I-cvi) is used evaluate the Content validity. I-cvi≥ 0.78 means the content validity is satisfactory.
  The Exploratory Factor Analysis (EFA) is used evaluate the Construct validity. The Kaiser-Mayer-Olkin (KMO) index (>0.6) is used to evaluate adaptability for factor analysis. Factor loading should >0.4.
  The Responsiveness analysis is used to evaluate the ability of this cognitive test that can reflect the change of cognitive function of the Interviewer during operation. Paired t-test can be used to compare whether the difference in score before and after is statistically significant. P value should < 0.05.

SECONDARY OUTCOMES:
PND (Perioperative neurocognitive disorders) | Baseline Test：1 day before operation, Second Test: Day 7 after operation
  PND is diagnosed by calculating the Z-score. The investigators get the score or accuracy and completion time of each test through the cognitive test network platform.
  Then Calculate Z-score: For each test, the mean practice effect is subtracted from the difference between preoperative and postoperative test scores; the result is then divided by the control group standard deviation to obtain a z-score. The z-scores of all tests in an individual patient are summarized and divided by the standard deviations for this sum of z-scores in the control subjects, creating a composite z-score.
  Cognitive decline is defined when two z-scores in individual tests or the composite z-score ≤-1.96.
  Perioperative neurocognitive disorders (PND) mainly refer to neurocognitive decline detected after surgery and anesthesia.